CLINICAL TRIAL: NCT04525248
Title: High Resection vs. Low Resection of Rectum in Laparoscopic Total Colectomy for Slow Transit Constipation
Brief Title: Resection Location of Rectum in Laparoscopic Surgery for Slow Transit Constipation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Minimally Invasive Surgery Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MISC-Constipation-Rectum
Record Dates: First submitted 2020-08-18; First posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Slow Transit; Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High resection (Active Comparator): Laparoscopic total colectomy + High resection of rectum
  Interventions: Procedure: Laparoscopic total colectomy + High resection of rectum
- Low resection (Experimental): Laparoscopic total colectomy + Low resection of rectum
  Interventions: Procedure: Laparoscopic total colectomy + low resection of rectum

INTERVENTIONS:
Procedure: Laparoscopic total colectomy + low resection of rectum — Laparoscopic total colectomy + low resection of rectum
  Arms: Low resection
Procedure: Laparoscopic total colectomy + High resection of rectum — Laparoscopic total colectomy + High resection of rectum
  Arms: High resection

SUMMARY:
Study the recurrence rate of constipation after laparoscopic total colectomy with high resection or low resection of rectum

DETAILED DESCRIPTION:
The investigators are going to study the recurrence rate of constipation after laparoscopic total colectomy with high resection or low resection of rectum. High resection is defined as resection at 12~15cm from anus and low resection as 6~8cm.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as constipation according to Rome IV criteria
* Diagnosed as slow transit constipation
* With more than 2 years' drug treatment or with outlet obstruction or with surgical history

Exclusion Criteria:

* Colon cancer
* History of colon, rectum, anus surgery
* With severe cardio, renal, neural disease
* Pregnant patients

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
1-year recurrence rate of constipation | 1 year
  1-year recurrence rate of constipation

SECONDARY OUTCOMES:
1-year rate of diarrhea | 1 year
  1-year rate of diarrhea
perioperative complications | 1 year
  perioperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Minhua Zheng, Study Chair — Shanghai MISC

IPD SHARING:
Plan to Share IPD: No